CLINICAL TRIAL: NCT03138044
Title: Long Term Outcome of Combined Ipsilateral Liver Lobe Devascularization and Alcohol Treatment (CILDAT) of the Large Hepatocellular Carcinoma (HCC)
Brief Title: Combined Ipsilateral Liver Lobe Devascularization and Alcohol Treatment of the Large Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The National Ribat University (Other)
Responsible Party: Principal Investigator, Osama Mohamed Elsanousi, General Surgeon, The National Ribat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS-003-17
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Ipsilateral Liver Lobe Devascularization; Alcohol Treatment; CILDAT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Combined Modality Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized and time series clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Treatment (Experimental): The Combined Treatment: patients undergo a surgical operation of ipsilateral liver lobe devascularization and four weeks later after the operation percutaneous alcohol injection sessions.
  Interventions: Procedure: Combined Treatment

INTERVENTIONS:
Procedure: Combined Treatment — This modality of palliative treatment includes initial surgical operation where arterial vascular supply of the tumor carrying liver lobe of the corresponding hepatic artery as well as the extrahepatic collateral arteries (EHCAs) feeding the large HCC (> 5 cms size) under general anesthesia. Four weeks after the operation the tumor is injeted (intralesionally and intravascularly) with absolute ethanol alcohol injections on regular weekly percutaneous sessions until the tumor become saturated and its vascularity rendered inactive.
  Other Names: CILDAT

SUMMARY:
Assessment of the long-term outcome of combined ipsilateral liver lobe devascularization (ILAD) and alcohol injection of the large hepatocellular carcinoma (HCC): single center non-randomized trial.

DETAILED DESCRIPTION:
Assessment of the overall (OS); one year; two years and three years' survival rates; the disease free survival (DFS) and the tumor response rate in the patients undergoing Combined Ipsilateral Liver Lobe Devascularization and Alcohol Treatment (CILDAT) of the Large HCC. This is a prospective non randomized trial carried out at the Ribat University Hospital between May 2017 to April 2020.

ELIGIBILITY:
Inclusion Criteria:

* Review and sign informed consent;
* Between 15 and 80 years of age at time of trial enrollment;
* Documented pathological and/or radiological diagnosis of hepatocellular carcinoma;
* Radiologically documented tumor size of > 5 centimeters;
* Radiologically documented liver cirrhosis.

Exclusion Criteria:

* American Anesthesia Association (ASA) Class IV or V and/or any contraindications to general anesthesia;
* Uncontrollable ascites;
* Deep persistent jaundice;
* Hepatic encephalopathy;
* Coagulopathy;
* Severe uncorrectable thrombocytopenia;
* Unable or unwilling to attend follow up visits and examinations;

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 3 years
  The percentage of patients who are still alive for three years after they started CILDAT for their large HCC.

SECONDARY OUTCOMES:
Disease free survival | 3 years
  Percentage of HCC patients who are alive and well (without a recurrence of their HCC) 3 years after CILDAT
Major complications' rate | 3 years
  Incidence of post CILDAT Clavien-Dindo comlicatins grade 3b or more.
Major toxicity rate | 3 years
  Incidence of post CILDAT Common Terminology Criteria for Adverse Events (CTCAE v4.03) grade
Tumor response rate | 3 years
  Mean percentage reduction in the sizes of the patients' tumors

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Elsanousi, MD, Principal Investigator — The National Ribat University
Locations (1):
- Ribat University Hospital, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elsanousi OM, Mohamed MA, Salim FH, Adam EA, Bedri S. Long-term outcome of novel combined surgical-injection treatment (COSIT) for large hepatocellular carcinoma: Stage 2A IDEAL prospective case series. Ann Med Surg (Lond). 2021 Nov 24;72:103098. doi: 10.1016/j.amsu.2021.103098. eCollection 2021 Dec. PMID 34888043